CLINICAL TRIAL: NCT03518892
Title: Assessing Dietary Requirements in Relation to Resting Metabolic Rate in Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 7333
Record Dates: First submitted 2018-04-11; First posted 2018-05-08 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Spinal Cord Injuries; Dietary Habits
Keywords: Resting Metabolic Rate
MeSH Terms: conditions — Spinal Cord Injuries; Feeding Behavior | interventions — Basal Metabolism; Body Composition; Nutrition Assessment

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Spinal Cord Injury Group: Body Composition, Resting Metabolic Rate, and dietary assessment
  Interventions: Diagnostic Test: Resting Metabolic Rate; Diagnostic Test: Body Composition; Behavioral: Dietary Assessment
- Healthy Controls: Body Composition, Resting Metabolic Rate, and dietary assessment
  Interventions: Diagnostic Test: Resting Metabolic Rate; Diagnostic Test: Body Composition; Behavioral: Dietary Assessment

INTERVENTIONS:
Diagnostic Test: Resting Metabolic Rate — 30 minute test to determine daily caloric needs
Diagnostic Test: Body Composition — Total Body DXA scan to determine fat mass, fat-free mass, and percent body fat
Behavioral: Dietary Assessment — Self administered dietary logs

SUMMARY:
Assess the relationship between body composition, metabolism, and dietary needs in people with spinal cord injury compared to their healthy controls that are age and sex matched.

DETAILED DESCRIPTION:
This study will quantify body composition and resting metabolic rate and then compare these parameters to results from a nutritional analysis. Participants will have two study visits that include physical exam, blood draws, resting metabolic rate, Dual Energy X-ray Absorptiometry (DXA) scan, and dietary assessments.

ELIGIBILITY:
Inclusion Criteria:

1. C4-L2 motor complete (AIS A & B) Spinal Cord injury for duration greater than 12 months.

4. <5% change in body in body weight over the past 12 months 5. Fluent in written and spoken English

Exclusion Criteria:

1. <22% body fat
2. Coronary artery disease
3. Type 1 diabetes mellitus, insulin-requiring Type 2 or untreated diabetes mellitus (fasting glucose>126 or HgbA1c>7.0)
4. Hypothyroidism, and/or renal disease
5. Decisional impairment
6. Prisoner

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Spinal Cord Injury subjects and healthy controls across central Pennsylvania.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Percentage of Body fat | Week 2
Fat Free Mass | Week 2
  lbs
Fat Mass | Week 2
  lbs
Resting Metabolic Rate | Week 2
Dietary Assessment Using Self-Reported Diary Questionaire | Week 2
  Dietary information will be collected from the participants using a self-reported food frequency diary questionnaire. The diary will log food, amount eaten, how it was prepared, and brand name of participant food intake at breakfast, lunch, snacks, and dinner.

CONTACTS AND LOCATIONS:
Overall Officials: David Gater, MD, PhD, MS, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No